CLINICAL TRIAL: NCT05992935
Title: A Phase 1/2, Randomized, Placebo-Controlled, Observer-Blind, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1403 and mRNA-1405, Multivalent Candidate Vaccines to Prevent Norovirus Acute Gastroenteritis in Healthy Adults 18 to 80 Years of Age
Brief Title: Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1403 and mRNA-1405 to Prevent Norovirus Acute Gastroenteritis in Healthy Adults 18 to 80 Years of Age
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1403/1405-P101
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Norovirus Acute Gastroenteritis
Keywords: mRNA-1403; mRNA-1405; Norovirus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Phase 1 Part: mRNA-1403 Dose Level 1 (Experimental): Participants will receive 2 intramuscular (IM) injections of mRNA-1403 at Dose Level 1.
  Interventions: Biological: mRNA-1403
- Phase 1 Part: mRNA-1403 Dose Level 2 (Experimental): Participants will receive 2 IM injections of mRNA-1403 at Dose Level 2.
  Interventions: Biological: mRNA-1403
- Phase 1 Part: mRNA-1403 Dose Level 3 (Experimental): Participants will receive 2 IM injections of mRNA-1403 at Dose Level 3.
  Interventions: Biological: mRNA-1403
- Phase 1 Part: mRNA-1403 Dose Level 4 Regimen 1 (Experimental): Participants will receive 2 IM injections of mRNA-1403 at Dose Level 4.
  Interventions: Biological: mRNA-1403
- Phase 1 Part: mRNA-1403 Dose Level 4 Regimen 2 (Experimental): Participants will receive 1 IM injection of mRNA-1403 at Dose Level 4 and 1 IM injection of study vaccine-matching placebo.
  Interventions: Biological: mRNA-1403; Biological: Placebo
- Phase 1 Part: mRNA-1405 Dose Level 1 (Experimental): Participants will receive 2 IM injections of mRNA-1405 at Dose Level 1.
  Interventions: Biological: mRNA-1405
- Phase 1 Part: mRNA-1405 Dose Level 2 (Experimental): Participants will receive 2 IM injections of mRNA-1405 at Dose Level 2.
  Interventions: Biological: mRNA-1405
- Phase 1 Part: mRNA-1405 Dose Level 3 (Experimental): Participants will receive 2 IM injections of mRNA-1405 at Dose Level 3.
  Interventions: Biological: mRNA-1405
- Phase 1 Part: mRNA-1405 Dose Level 4 Regimen 1 (Experimental): Participants will receive 2 IM injections of mRNA-1405 at Dose Level 4.
  Interventions: Biological: mRNA-1405
- Phase 1 Part: mRNA-1405 Dose Level 4 Regimen 2 (Experimental): Participants will receive 1 IM injections of mRNA-1405 at Dose Level 4 and 1 IM injection of study vaccine-matching placebo.
  Interventions: Biological: mRNA-1405; Biological: Placebo
- Phase 1 Part: Placebo (Placebo Comparator): Participants will receive 2 IM injections of study vaccine-matching placebo.
  Interventions: Biological: Placebo
- Phase 2 Part: mRNA-1403 Dose Level 1 (Experimental): Participants will receive 1 IM injection of mRNA-1403 at Dose Level 1.
  Interventions: Biological: mRNA-1403
- Phase 2 Part: mRNA-1403 Dose Level 2 (Experimental): Participants will receive 1 IM injection of mRNA-1403 at Dose Level 2 and if participating in the booster extension will receive a second dose of mRNA-1403 at Dose Level 3 or study vaccine-matching placebo 12-15 months after first dose.
  Interventions: Biological: mRNA-1403; Biological: Placebo
- Phase 2 Part: mRNA-1403 Dose Level 3 (Experimental): Participants will receive 1 IM injection of mRNA-1403 at Dose Level 3 and if participating in the booster extension will receive a second dose of mRNA-1403 at Dose Level 3 or study vaccine-matching placebo 12-15 months after first dose.
  Interventions: Biological: mRNA-1403; Biological: Placebo
- Phase 2 Part: Placebo (Placebo Comparator): Participants will receive 1 IM injection of study vaccine-matching placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1403 — Sterile liquid for injection
  Arms: Phase 1 Part: mRNA-1403 Dose Level 1; Phase 1 Part: mRNA-1403 Dose Level 2; Phase 1 Part: mRNA-1403 Dose Level 3; Phase 1 Part: mRNA-1403 Dose Level 4 Regimen 1; Phase 1 Part: mRNA-1403 Dose Level 4 Regimen 2; Phase 2 Part: mRNA-1403 Dose Level 1; Phase 2 Part: mRNA-1403 Dose Level 2; Phase 2 Part: mRNA-1403 Dose Level 3
Biological: mRNA-1405 — Sterile liquid for injection
  Arms: Phase 1 Part: mRNA-1405 Dose Level 1; Phase 1 Part: mRNA-1405 Dose Level 2; Phase 1 Part: mRNA-1405 Dose Level 3; Phase 1 Part: mRNA-1405 Dose Level 4 Regimen 1; Phase 1 Part: mRNA-1405 Dose Level 4 Regimen 2
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Phase 1 Part: Placebo; Phase 1 Part: mRNA-1403 Dose Level 4 Regimen 2; Phase 1 Part: mRNA-1405 Dose Level 4 Regimen 2; Phase 2 Part: Placebo; Phase 2 Part: mRNA-1403 Dose Level 2; Phase 2 Part: mRNA-1403 Dose Level 3

SUMMARY:
The purpose of the Phase 1 Part of this study is to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1403 and mRNA-1405 in healthy adult participants 18 to 49 years of age and 60 to 80 years of age. The purpose of the Phase 2 Part of the study is to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1403 in healthy adult participants 18 to 80 years of age.

ELIGIBILITY:
Key Inclusion Criteria:

* Phase 1 Part: Adults 18 to 49 years of age at the time of consent or adults 60 to 80 years of age at the time of consent.
* Phase 2 Part: Adults 18 to 80 years of age at the time of consent.
* Body mass index of 18 to 39 kilogram/meter^2 (inclusive) at the Screening Visit (relevant only for the base period of Phase 1 and Phase 2).
* Participants assigned female at birth are eligible to participate if they are not pregnant or breast/chest/body feeding.
* A person of childbearing potential is using a highly effective contraceptive method.
* Participant has provided written informed consent for participation in this study.

Key Exclusion Criteria:

* Is acutely ill or febrile (temperature ≥38.0°C [100.4°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Phase 2 Part booster extension period: acute disease or febrile 72 hours prior to or on Day 365.
* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Has a medical, psychiatric, or occupational condition, including reported history of substance abuse, which may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment.
* Has a current or previous diagnosis of immunosuppressive condition, to include human immunodeficiency virus, or immune-mediated (autoimmune) disease that requires immunosuppressive therapies.

(drugs or biologics). The use of topical corticosteroids or other immunosuppressive agents (for example, topical calcineurin inhibitor) may be eligible for participation at the discretion of the Investigator.

* History of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine or intervention that includes one or more of the same components contained in the study vaccine.
* Phase 1 Part and Phase 2 Part base period: Any history of myocarditis or pericarditis.
* Phase 2 Part booster extension period: Any history of myocarditis, pericarditis, or Guillain-Barré Syndrome.
* Coagulopathy or bleeding disorder considered a contraindication to IM injection or phlebotomy.
* Dermatologic conditions that could affect local solicited AR assessments (for example, tattoos, psoriasis patches affecting skin over the deltoid areas).
* Has received systemic immunosuppressive therapies (drugs or biologics) for >14 days in total within 6 months prior to Screening or Day 365 (Phase 2 Part booster extension period only) (for corticosteroids ≥10 mg/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study. Inhaled, nasal, intra-articular, and topical steroids are allowed.
* Has received or plans to receive any licensed/authorized vaccine (to include severe acute respiratory syndrome-related coronavirus-2 vaccine) ≤28 days prior to or within 28 days after each study intervention, with the exception of influenza vaccines, which may be given 14 days before or after receipt of a study intervention.
* Has received systemic immunoglobulins or blood products within 3 months prior to Screening or Day 365 (Phase 2 Part booster extension period only) or plans for receipt during the study.
* Has donated protocol-specified volume of blood products within protocol-specified timeframe.
* Participated or plans to participate in an interventional clinical study within protocol-specified timeframe.
* Phase 2 Part: Individuals who are participating/have participated in the Phase 1 part of the study are excluded.
* Phase 1 Part: Any individual with laboratory abnormalities achieving thresholds defined in the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1285 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to a maximum of Day 36 (7 days after each study injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to a maximum of Day 57 (28 days after each study injection)
Number of Participants with Medically Attended AEs (MAAEs) | Day 1 up to a maximum of Day 197
Number of Participants with Any Serious Adverse Events (SAEs), AEs Leading to Withdrawal From Study/Discontinuation of Study Vaccine, and Adverse Events of Special Interest (AESIs) | Day 1 up to a maximum of Day 365

SECONDARY OUTCOMES:
Geometric Mean Titers (GMT) of Histo-blood Group Antigen (HBGA)-blocking Antibodies Against Vaccine-matched Norovirus (NoV) Genotypes | Phase 1: Days 1, 29, and 57; Phase 2: Days 1, 29, 365, and 393
Geometric Mean Fold Rise (GMFR) of HBGA-blocking Antibodies Titers | Phase 1: Days 1, 29, and 57; Phase 2: Days 1, 29, 365, and 393
Percentage of Participants with Seroresponse Based on HBGA-blocking Antibody Titers | Phase 1: Days 29, and 57; Phase 2: Days 29 and 393
Geometric Mean Concentration (GMC) of Binding Antibody (bAb) Against Vaccine-matched NoV Genotypes | Days 1, 29, and 57
GMFR of bAb Levels | Days 1, 29, and 57
Percentage of Participants with Seroresponse Based on bAb Levels | Days 29 and 57

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - ARK Clinical Research, LLC, Long Beach, California
  - Tekton Research, Inc - Longmont Center, Longmont, Colorado
  - Research Centers of America, Hollywood, Florida
  - Accel Research Sites Network, Decatur, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Optimal Research, Peoria, Illinois
  - Velocity Clinical Research, Sioux City, Iowa
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - Velocity Clinical Research, Rockville, Maryland
  - Velocity Clinical Research, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Rochester Clinical Research, Inc, Rochester, New York
  - Epic Medical Research, LLC, Red Oak, Texas
  - JBR Clinical Research, Salt Lake City, Utah